CLINICAL TRIAL: NCT03123926
Title: Spontaneous Preterm Birth Marker Test (SPBMT): Preterm Prediction Prospective Study
Brief Title: Spontaneous Preterm Birth Marker Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sprim Advanced Life Sciences (Other)
Collaborators: BABYNOSTICS (Unknown)
Responsible Party: Sponsor
Other Study IDs: BAB-0316
Record Dates: First submitted 2017-02-20; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Preterm Delivery
Keywords: spontaneous preterm birth; lipids; biomarkers
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva, cervicovaginal fluid, serum and dried blood spot
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prediction of preterm birth is beneficial because it initiates early treatment to minimize risk. It defines a population at risk to provide particular treatment and may lead us to a better understanding the mechanisms of preterm birth. The understanding of the mechanisms and etiology consequently leads to the possibility of early intervention and effective management aiming at preventing preterm birth. Five most common interventions for preventing and treating preterm birth are antibiotics, cervical cerclage, bed rest, progesterone, and tocolytic therapy. However, there are insufficient evidence showing the efficacy of cerclage and bed rest; antibiotics may only delay but not prevent the preterm birth; the use of certain tocolytics needs to be considered against the possible adverse effects. The early detection of pregnant women with high risk for preterm delivery would be the ideal solution to prevent preterm birth. However, to date, there is inadequate literature and little knowledge of diagnosis, treatment, prevention and prediction of preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy women aged ≥ 18 years with pregnancy at 24 to 28 weeks of gestation.

Exclusion Criteria:

* Subjects with any conditions or diseases that investigator considers it is not appropriate to enter the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy women
Study Population: Estimated 600 symptomatic women aged ≥ 18 years with pregnancy at 24 to 28 weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cervical length | 6-12 months
  Cervical length <15, 20, 25 mm
Biomarkers (serum) | 6-12 months
  subjects with feral fibronectin ≥50 ng/mL, >10 mg/L of cervical phIGFBP1; elevated Interleukin-6 as compared to term birth; significantly present of other biomarkers.
Lipid analysis (serum and DBS) | 6-12 months
  Lipid profiles of preterm birth compared to term birth.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Diosdado V., MD, Principal Investigator — MD
Locations (1):
- The Perinatal Association of the Philippines, Quezon, Brgy Malaya, Philippines